CLINICAL TRIAL: NCT05850247
Title: Plaque and Brain Inflammation in Symptomatic Carotid Stenosis: Role of the Ficolin-2
Acronym: STATEMENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0403; 2023-504573-20 (EudraCT Number)
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: CAROTID STENOSIS
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]DPA-714 PET/MRI (Experimental)
  Interventions: Drug: [18F]DPA-714 PET/MRI

INTERVENTIONS:
Drug: [18F]DPA-714 PET/MRI — To assess the association between plasma ficolin-2 levels and plaque and brain inflammation assessed by [18F]DPA-714 PET/MRI in patients managed for transient ischaemic attack or ischaemic stroke related to carotid stenosis.
  PET/MRI of the brain and carotid plaque with [18F]DPA-714 and gadolinium infusion will be performed at day 5.

SUMMARY:
Carotid artery stenosis is observed in about 3% of ≥ 60 years subjects and accounts for around 10-20% of all ischemic strokes. Beyond the degree of stenosis, plaque composition affects the risk of ischemic stroke. Identification of patients with vulnerable plaques at higher risk of stroke who might benefit from carotid revascularization is crucial.

A growing body of evidence suggests that the lectin pathway of the complement system, and especially the ficolin-2, is involved in atherosclerosis. It has been hypothesized that circulating levels of ficolin-2 increase during chronic inflammatory conditions (i.e. growing atherosclerotic plaque) whereas they fall during sub-acute or acute inflammatory conditions (i.e. plaque rupture and acute ischemic stroke) because of consumption (binding to targets). Therefore, ficolin-2 has been proposed as a biomarker informing on the specific state of the plaque. However, in acute ischemic stroke due to carotid stenosis, both plaque rupture and stroke injury contribute to lectin pathway activation, thus affecting circulating levels of ficolin-2. Until now, the relative contribution of plaque and brain inflammation on circulating levels of ficolin-2 has not been documented.

In the present study the investigators aim to assess the association between circulating levels of ficolin-2 and carotid and brain inflammation on [18F]DPA-714 positron emission tomography (PET)/MRI in patients with transient ischemic attack or acute ischemic stroke due to carotid stenosis. For that purpose, the investigators intend to include 30 patients with transient ischemic attack or acute ischemic stroke due to ≥ 50%. carotid stenosis. Each patient will have a measure of plasmatic level of ficolin-2 as well a [18F]DPA-714 PET/MRI to quantify the fixation of the radiotracer on carotid and brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or over,
* Signed written informed consent before any study specific intervention,
* Probable ipsilateral transient ischemic attack (TIA - which involve a focal speech/language, motor or visual deficit referable to the distribution of a carotid artery and lasting less than 48 hours from the onset) OR retinal artery occlusion ≤ 48h OR ischemic stroke ≤ 48h from the onset,
* Atherosclerotic carotid stenosis between 50% and 99% (NASCET method), as confirmed by one of the imaging examinations (among: Doppler ultrasound, MR angiography, CT angiography, catheter angiography) performed after index TIA or ischemic stroke
* No other identified cause of TIA, ischemic stroke or retinal artery occlusion,

Exclusion Criteria:

* Patients with inflammatory or autoimmune disease, hepatocellular insufficiency, acute or chronic infection, active malignancy, myocardial infarction or major surgery within the previous 30 days of index hospitalization according to the investigator,
* Patients with severe renal insufficiency (estimated GFR < 30 ml/min at inclusion or known dialysis),
* Patients with contraindication to MRI (agitation, claustrophobia, pacemaker, metallic (ferromagnetic) body, a known allergy to gadolinium) according to the investigator's judgment,
* Patients with modified Rankin score greater than 3,
* Patients currently enrolled in another clinical trial including investigational medicinal products,
* Female patient who is pregnant or lactating, or is of child-bearing and who did not agree to use highly effective methods of birth control throughout the study,
* Patient without health coverage,
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between: - Plasma levels of ficolin-2 at day 5 in ng/ml, - Metabolic data on [18F]DPA-714 PET/MRI | day 5
  To assess the association between circulating levels of ficolin-2 and carotid and brain inflammation on [18F]DPA-714 PET/MRI in patients with transient ischemic attack or acute ischemic stroke due to carotid stenosis

SECONDARY OUTCOMES:
Correlation between plasma levels of ficolin-2 at day 5 in ng/mL with morphological data of the brain and carotid plaque assessed by MRI | day 5
  To assess if plasma levels of ficolin-2 in patients with TIA or acute ischemic stroke due to carotid stenosis correlate with:
  1. morphological data:
  * of the plaque: presence of intraplaque hemorrhage, lipid-rich necrotic core, thinning/rupture of the fibrous cap on carotid plaque MRI
  * of the brain: infarct size, presence of hemorrhagic transformation, blood-brain barrier leakage
Correlation between plasma levels of ficolin-2 at day 5 in ng/mL with morphological data of the brain and carotid plaque assessed by MRI | day 15
  To assess if plasma levels of ficolin-2 in patients with TIA or acute ischemic stroke due to carotid stenosis correlate with:
  - histological data of the retrieved plaque: hemorrhagic content, lipid core, cholesterol cleft areas, ratio between thickness of tunica media and total thickness of tunica, rupture, intraplaque deposition of ficolin-2, macrophages and neutrophils infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Laura MECHTOUFF, Principal Investigator — Service de Neurologie vasculaire / CarMeN U1060 INSERM
Locations (1):
- Service de Neurologie vasculaire / CarMeN U1060 INSERM Hôpital Neurologique Pierre Wertheimer - GHE, Bron, France